CLINICAL TRIAL: NCT00416052
Title: Relation Between Bone Mineral Density and the Regulation of Mineral Metabolism in Renal Stone Formers
Brief Title: Relation Between Bone Density and the Regulation of Mineral Metabolism in Renal Stone Formers
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Andreas Pasch, Department of Nephrology and Hypertension, Inselspital, University Hospital Bern
Other Study IDs: BE001
Record Dates: First submitted 2006-12-26; First posted 2006-12-27 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Calcium Nephrolithiasis
Keywords: calcium; calciuria; PTH; 1,25-vitamin D; Calcitriol; bone mineral density; osteodensitometry

STUDY DESIGN:
Observational Model: Case-Only

SUMMARY:
Accumulating evidence indicated that renal calcium stone formers often exhibit a low bone density. Therefore we want to test the hypothesis, that the mineral (calcium) metabolism is differently regulated in calcium stone formers with low as opposed to high bone density.

DETAILED DESCRIPTION:
There is epidemiological evidence associating renal calcium stones and decreased bone mineral density (BMD). The decreased BMD in calcium stone formers is linked to hypercalciuria and both subtypes, fasting as well as absorptive hypercalciuria are associated with a diminished BMD. Higher 1,25-vitamin D plasma concentrations and lower PTH levels are encountered under free-choice diet conditions in patients diagnosed with absorptive and fasting hypercalciuria when compared to normocalciuric stone formers. Reports studying the BMD of stone formers and its link with mineral metabolism variables and urinary calcium excretion under different calcium intakes are rare.

We hypothesize now that PTH and 1,25-vitamin D change differently when calcium stone formers with high, intermediate and low BMD are challenged by a low calcium diet.

ELIGIBILITY:
Inclusion Criteria:

* passage of at least one calcium containing kidney stone

Exclusion Criteria:

* established cause of calcium stone formation (sarcoidosis, primary hyperparathyroidism etc.)
* creatinine clearance < 60 ml/min
* urinary tract infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recurrent renal calcium stone formers
Sampling Method: Non-Probability Sample
Enrollment: 90
Dates: Start 2004-03; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Felix J Frey, MD, Study Director — University of Bern
Locations (1):
- Dept. Nephrology & Hypertension, Univ. Hospital Bern, Bern, Switzerland